CLINICAL TRIAL: NCT02710227
Title: Sleep Timing and Circadian Preferences in A Sample of Egyptian Patients With Hepatic Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, MD liver diseases, Tanta University
Organization: Tanta University (Other)
Other Study IDs: Sleep Patterns in cirrhotics
Record Dates: First submitted 2016-03-09; First posted 2016-03-16 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- liver cirrhosis: Sleep quality, sleep timing parameters and circadian preference were evaluated using (PSQI), (STQ).
  Interventions: Other: (PSQI), (STQ).
- control: Sleep quality, sleep timing parameters and circadian preference were evaluated using (PSQI), (STQ).
  Interventions: Other: (PSQI), (STQ).

INTERVENTIONS:
Other: (PSQI), (STQ). — Sleep quality, sleep timing parameters and circadian preference were evaluated using (PSQI), (STQ).

SUMMARY:
Individuals with hepatic cirrhosis (n=50) and healthy controls (n=30) were recruited. Sleep quality, sleep timing parameters and circadian preference were evaluated using the Pittsburgh Sleep Quality Index (PSQI), Sleep Timing Questionnaire (STQ) and The Composite Scale for Morningness (CSM) respectively

DETAILED DESCRIPTION:
Cirrhosis of the liver is a chronic, diffuse, degenerative disease in which the parenchyma deteriorates, the lobules are infiltrated with fat and structurally altered, dense perilobular connective tissue forms and often areas of regeneration develop. These regeneration nodules have a reduced blood supply resulting in impaired liver function [1] and [2]. Factors that are taken into account to determine the severity of cirrhosis include serum albumin, prothrombin concentration, serum bilirubin, ascites and encephalopathy. A point system known as the Child's-pough-Turcotte score has been designed to determine the severity of cirrhosis. Depending on the total score, patients are classified as class A (early cirrhosis) through class C (advanced cirrhosis) [3].

A disturbance of sleep is recognized as one of the early signs of hepatic encephalopathy. Reversal of sleep rhythm, drowziness and lethargy are classic signs of this disease. Sleep disturbance and excessive daytime somnolence are common in patients with cirrhosis. It was estimated that up to 70% of individuals with cirrhosis (regardless of etiology) experience sleep disturbances [4]. Difficulty falling asleep and a shift in sleep schedule toward the latter part of the night, which might be result in daytime sleepiness, are commonly reported findings in patients with hepatic cirrhosis without encephalopathy [4].

Individuals with hepatic cirrhosis (n=50) and healthy controls (n=30) were recruited. Sleep quality, sleep timing parameters and circadian preference were evaluated using the Pittsburgh Sleep Quality Index (PSQI), Sleep Timing Questionnaire (STQ) and The Composite Scale for Morningness (CSM) respectively

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis
* controls

Exclusion Criteria:

* HCC

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with hepatic cirrhosis (n=50) and healthy controls (n=30) were recruited.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of individuals with sleep disturbances | 1 year
  Number of individuals with sleep disturbances among cirrhotics

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed yousef, MD, Principal Investigator — Hepatology and gastroenterology dept.-Tanta; Mohamed seleem, MD, Study Director — Neuropsychiatry dept.- Tanta; Sherief Abd-Elsalam, MD, Study Director — Hepatology and gastroenterology dept.-Tanta; Mohamed Elhendawy, MD, Study Chair — Hepatology and gastroenterology dept.-Tanta; Sabry Abou saif, MD, Study Chair — Hepatology and gastroenterology dept.-Tanta; Abdelrahman Kobtan, MD, Study Chair — Hepatology and gastroenterology dept.-Tanta
Locations (1):
- Tanta university - faculty of medicine, Tanta, Elgharbia, Egypt

IPD SHARING:
Plan to Share IPD: No